CLINICAL TRIAL: NCT01410201
Title: Dexamethasone Intravitreal Implant After Vitrectomy for Idiopathic Epiretinal Membrane
Brief Title: Dexamethasone Intravitreal Implant After Vitrectomy For Epiretinal Membrane
Acronym: OZURDEX2
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recruitment not met
Sponsor: Barnes Retina Institute (Other)
Collaborators: Allergan (Industry)
Responsible Party: Principal Investigator, Rhonda Weeks, Gaurav K. Shah, MD, Barnes Retina Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OZURDEX ERM
Record Dates: First submitted 2011-07-19; First posted 2011-08-05 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-07

CONDITIONS: Epiretinal Membrane; Macular Edema
Keywords: Epiretinal Membrane; Macular Edema; Dexamethasone Intravitreal Implant (Ozurdex); Pars Plana Vitrectomy
MeSH Terms: conditions — Epiretinal Membrane; Macular Edema | interventions — Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PPV + MP + DEX (Experimental): Patients will undergo pars plana vitrectomy, membrane peel, and concomitant Ozurdex implant (0.7 mg dose).
  Interventions: Drug: Dexamethasone Intravitreal Implant
- PPV + MP (Active Comparator): Patients will undergo pars plana vitrectomy with membrane peel, without Ozurdex implant.
  Interventions: Drug: Dexamethasone Intravitreal Implant

INTERVENTIONS:
Drug: Dexamethasone Intravitreal Implant — Half of the study participants (15 out of 30) will receive one - Dexamethasone Intravitreal Implant 0.7 mg.
  Other Names: Pars Plana Vitrectomy; Membrane Peel; Dexamethasone Intravitreal Implant (Ozurdex)

SUMMARY:
The purpose of this study is to evaluate the effect of dexamethasone intravitreal implant (Ozurdex) in combination with pars plana vitrectomy and membrane peeling for idiopathic epiretinal membrane (ERM).

DETAILED DESCRIPTION:
Pars plana vitrectomy with membrane peeling has been used for years to successfully to treat ERM (epiretinal membrane). However, despite successful surgery, approximately 10-30% of patients may not experience any improvement in visual acuity (ref. 1-7). Macular causes of unsatisfactory visual outcome following vitrectomy include persistent macular edema and reoccurrence of epiretinal membrane (ref. 1-7). Concomitant administration of intravitreal corticosteroids (triamcinolone acetonide) after pars plana vitrectomy and membrane peeling for epiretinal membrane has been reported to speed up and improve the anatomic and functional outcome (ref 8). Given that intravitreal triamcinolone has been reported to last approximately 113 days ina post-vitrectomy eye (ref. 9); the investigators postulate that a longer-acting corticosteroid such as Ozurdex could not only have the benefits of improved anatomic and functional outcomes, but also a longer sustained effect.

ELIGIBILITY:
Inclusion Criteria:

* Patients with idiopathic epiretinal membrane
* Preoperative visual acuity of snellen equivalent 20/32 or worse

Exclusion Criteria:

* History or presence of any of the following:
* uveitis
* macular hole
* previous vitreoretinal surgery
* any other retinal pathology that could affect anatomic or functional results
* Age Related Macular Degeneration
* Diabetic Retinopathy
* Diabetic Macular Edema
* Retinal Vein Occlusion
* Pre-existing Macular Disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2011-08; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Changes in best corrected visual acuity | 6 months
  At all study visits:
  ETDRS visual acuity will be measured visit excluding post op day 1 (snellen visual acuity will be measured).
  Intraocular pressure (IOP) will be checked. Spectral Domain Optical Coherence Tomography (OCT). Dilated fundus exam.
  At Pre Op, Post Op Week 4, 8, 12, 16, 20 and 24 visits:
  ETDRS visual acuity will be measured. IOP check. Spectral Domain OCT. Fundus photography. Fundus Autofluorescence (AF). Fluorescein Angiography (FA). Dilated Fundus exam.

SECONDARY OUTCOMES:
Incidence of persistent macular edema on Central OCT thickness in treatment (PPV + MP + DEX) versus non-treatment (PPV + MP) groups | 6 months
  At all visits: ETDRS visual acuity will be measured except post op day 1 (snellen visual acuity will be measured) Intraocular pressure (IOP) will be checked Spectral Domain Optical Coherence Tomography (OCT) Dilated fundus exam
  At Pre Op, Post Op Week 4, 8, 12, 16, 20, and 24:
  ETDRS visual acuity will be measured IOP will be checked Spectral Domain OCT Fundus Photography Fundus Auto Fluorescence (AF) Fluorescein Angiography (FA) Dilated Fundus exam

CONTACTS AND LOCATIONS:
Overall Officials: Gaurav K Shah, MD, Principal Investigator — Retina Institute
Locations (3):
- United States (3):
  - St. Lukes Hospital, Chesterfield, Missouri
  - St. Louis Eye Surgery and Laser Center, St Louis, Missouri
  - The Retina Institute, St Louis, Missouri

REFERENCES:
- [Background] Smiddy WE, Michels RG, Green WR. Morphology, pathology, and surgery of idiopathic vitreoretinal macular disorders. A review. Retina. 1990;10(4):288-96. doi: 10.1097/00006982-199010000-00012. PMID 2089546
- [Background] de Bustros S, Thompson JT, Michels RG, Rice TA, Glaser BM. Vitrectomy for idiopathic epiretinal membranes causing macular pucker. Br J Ophthalmol. 1988 Sep;72(9):692-5. doi: 10.1136/bjo.72.9.692. PMID 3179258
- [Background] Michels RG. Vitrectomy for macular pucker. Ophthalmology. 1984 Nov;91(11):1384-8. doi: 10.1016/s0161-6420(84)34136-7. PMID 6514308
- [Background] McDonald HR, Verre WP, Aaberg TM. Surgical management of idiopathic epiretinal membranes. Ophthalmology. 1986 Jul;93(7):978-83. doi: 10.1016/s0161-6420(86)33635-2. PMID 3763143
- [Background] Schadlu R, Tehrani S, Shah GK, Prasad AG. Long-term follow-up results of ilm peeling during vitrectomy surgery for premacular fibrosis. Retina. 2008 Jun;28(6):853-7. doi: 10.1097/IAE.0b013e3181631962. PMID 18536602
- [Background] Koerner F, Garweg J. Vitrectomy for macular pucker and vitreomacular traction syndrome. Doc Ophthalmol. 1999;97(3-4):449-58. doi: 10.1023/a:1002412323399. PMID 10896363
- [Background] Massin P, Allouch C, Haouchine B, Metge F, Paques M, Tangui L, Erginay A, Gaudric A. Optical coherence tomography of idiopathic macular epiretinal membranes before and after surgery. Am J Ophthalmol. 2000 Dec;130(6):732-9. doi: 10.1016/s0002-9394(00)00574-2. PMID 11124291
- [Background] Konstantinidis L, Berguiga M, Beknazar E, Wolfensberger TJ. Anatomic and functional outcome after 23-gauge vitrectomy, peeling, and intravitreal triamcinolone for idiopathic macular epiretinal membrane. Retina. 2009 Sep;29(8):1119-27. doi: 10.1097/IAE.0b013e3181ac23da. PMID 19734764
- [Background] Kosobucki BR, Freeman WR, Cheng L. Photographic estimation of the duration of high dose intravitreal triamcinolone in the vitrectomised eye. Br J Ophthalmol. 2006 Jun;90(6):705-8. doi: 10.1136/bjo.2005.088278. Epub 2006 Mar 10. PMID 16531422